CLINICAL TRIAL: NCT01924065
Title: Does Cardioversion of Atrial Fibrillation Increase the Risk of Stroke and Silent Cerebrovascular Thromboembolism? Comparison of the Two Cardioversion Methods
Brief Title: Risk of Stroke and Silent Cerebrovascular Thromboembolism After Cardioversion of Atrial Fibrillation
Acronym: AFTER-CV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mehmet Ozaydin, MD, MD, Professor in Cardiology, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ozaydin291
Record Dates: First submitted 2013-08-07; First posted 2013-08-16 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation; Cardioversion; Cerebrovascular Stroke
Keywords: Atrial fibrillation, conversion, stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Electric Countershock; Anticoagulants

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transesophageal Echocardiography group (Active Comparator): This arm includes the patients with atrial fibrillation who undergo transesophageal echocardiography-guided cardioversion
  Interventions: Procedure: Cardioversion
- Oral anticoagulant Group (Active Comparator): This arm includes the patients with atrial fibrillation who take warfarin or new oral anticoagulant agents three weeks before electrical cardioversion.
  Interventions: Procedure: Cardioversion; Drug: Oral Anticoagulant

INTERVENTIONS:
Procedure: Cardioversion — Electrical cardioversion
Drug: Oral Anticoagulant — warfarin, dabigatran etexilate, rivaroxaban, apixaban, edoxaban usage
  Arms: Oral anticoagulant Group

SUMMARY:
Patients with atrial fibrillation undergoing cardioversion will be randomized to undergo transesophageal echocardiography or they will receive warfarin for 3 weeks with an international normalized ratio (INR) value between 2.0-3.0. Those who do not want to use warfarin will be given an approved new oral anticoagulant agent instead of warfarin for 3 weeks.

If thrombus is detected in left atrium or in left atrial appendage, no cardioversion will be performed. Other patients in the both groups will undergo electrical cardioversion. After the procedures all the patients will be given oral anticoagulant for at least 4 Weeks. All patients will have neurological examination and diffusion magnetic resonance imaging (MRI) at baseline and at postprocedural 7th day. Clinical and subclinical cerebral thromboembolic events detected by diffusion MRI will be recorded. Any bleeding events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the age of more than 18 years who are planned to undergo electrical or medical cardioversion

Exclusion Criteria:

* Urgent cardioversion
* Patients who have implanted pace-makers or other metal devices
* Claustrophobia
* Hematological disorders disabling patients to receive anticoagulant agents
* Atrial fibrillation secondary to temporary causes.
* Serious rheumatic heart valve disease
* Hyperthyroidism
* History of malignancy
* Left atrium diameter > 55 mm
* Ejection fraction < 0.25

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-08; Primary Completion 2017-08 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ozaydin, Professor,MD, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Mediterranean Region, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transesophageal Echocardiography Group | Oral Anticoagulant Group
Started | 56 | 56
Completed | 56 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transesophageal Echocardiography Group | Oral Anticoagulant Group | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] — higher values represent worse outcome
  years | 61 (10.5) | 60 (12.1) | 60.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 33 | 33 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 56 | 56 | 112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 56 | 56 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 56 | 56 | 112
Hypertension [Count of Participants; unit: Participants] | 27 | 27 | 54
Diabetes mellitus [Count of Participants; unit: Participants] | 17 | 12 | 29
Coronary artery disease [Count of Participants; unit: Participants] | 10 | 10 | 20
Heart rate [Mean (Standard Deviation); unit: Beats per minute] — higher values represent worse outcome
  Beats per minute | 104.5 (23.9) | 98.3 (23) | 101.5 (23.6)
Left atrial diameter [Mean (Standard Deviation); unit: mm] — higher values represent worse outcome
  mm | 41 (3.7) | 42.1 (3.4) | 41.6 (3.6)
Ejection fraction [Mean (Standard Deviation); unit: percent] — higher values represent better outcome
  percent | 61.3 (6.2) | 60 (6) | 60.5 (6.1)
Type of atrial fibrillation [Count of Participants; unit: Participants]
  Paroxysmal | 37 | 36 | 73
  Persistent | 19 | 20 | 39
Duration of atrial fibrillation [Median (Full Range); unit: day] — higher values represent worse outcome
  day | 3.5 [2 to 1825] | 4 [2 to 1095] | 4 [2 to 1825]
Beta blocker [Count of Participants; unit: Participants] | 19 | 33 | 52
Calcium channel blocker [Count of Participants; unit: Participants] | 11 | 9 | 20
Amiodarone [Count of Participants; unit: Participants] | 0 | 1 | 1
Propafenone [Count of Participants; unit: Participants] | 3 | 3 | 6
Acetylsalicylic acid [Count of Participants; unit: Participants] | 17 | 15 | 32
Clopidogrel [Count of Participants; unit: Participants] | 4 | 3 | 7
Angiotensin converting enzyme inhibitor, Angiotensin receptor blocker [Count of Participants; unit: Participants] | 20 | 20 | 40
Spironolactone [Count of Participants; unit: Participants] | 2 | 5 | 7
Congestive heart failure, Hypertension, Age 2, Diabetes, Stroke 2, Vascular, Sex Category Score [Mean (Standard Deviation); unit: units on a scale] — Congestive heart failure, Hypertension, Age 2, Diabetes, Stroke 2, Vascular, Sex Category (CHA2DS2-VASc) Score ranges from score 0 (lowest stroke risk) to 9 (highest stroke risk). The total score is provided; subscales are summed to compute a total score; higher values represent worse outcome
  units on a scale | 1.44 (1.11) | 1.62 (1.05) | 1.53 (1.08)
Hypertension,Abnormal liver/renal function, Stroke, Bleeding, LabileINR, Elderly, Drug/alcohol Score [Mean (Standard Deviation); unit: units on a scale] — Hypertension,Abnormal liver/renal function, Stroke, Bleeding, LabileINR, Elderly, Drug/alcohol (HAS-BLED) Score ranges from score 0 (lowest bleeding risk) to 9 (highest bleeding risk). Total score is provided; subscales are summed to compute a total score; higher values represent worse outcome
  units on a scale | 0.41 (0.59) | 0.39 (0.62) | 0.4 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Combined Clinical Thromboembolic or Hemorrhagic Event, Death or Silent Cerebral Thromboemboli
Description: Clinical events during 2 years follow-up or silent cerebral thromboemboli detected by diffusion magnetic resonance imaging at 1 week post-cardioversion
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Transesophageal Echocardiography Group | Oral Anticoagulant Group
Number analyzed (Participants) | 56 | 56
Participants | 9 | 11

2. Primary Outcome: Efficacy Clinical End-point
Description: Any Clinical Thromboembolic Event, Death or Silent Cerebral Thromboemboli
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Transesophageal Echocardiography Group | Oral Anticoagulant Group
Number analyzed (Participants) | 56 | 56
Participants | 7 | 9

3. Primary Outcome: Ischemic Stroke/Transient Ischemic Attack
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Transesophageal Echocardiography Group | Oral Anticoagulant Group
Number analyzed (Participants) | 56 | 56
Participants | 7 | 4

4. Primary Outcome: Acute Ischemia in MRI
Description: Development of acute silent cerebral ischemia detected by MRI
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Transesophageal Echocardiography Group | Oral Anticoagulant Group
Number analyzed (Participants) | 56 | 56
Participants | 2 | 4

5. Primary Outcome: Mortality
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Transesophageal Echocardiography Group | Oral Anticoagulant Group
Number analyzed (Participants) | 56 | 56
Participants | 3 | 2

6. Primary Outcome: Hemorrhagic Stroke
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Transesophageal Echocardiography Group | Oral Anticoagulant Group
Number analyzed (Participants) | 56 | 56
Participants | 1 | 2

7. Primary Outcome: Gastrointestinal Bleeding
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Transesophageal Echocardiography Group | Oral Anticoagulant Group
Number analyzed (Participants) | 56 | 56
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Oral Anticoagulation Group: This arm includes the patients with atrial fibrillation who take warfarin or new oral anticoagulant agents three weeks before electrical cardioversion.
  Cardioversion: Electrical cardioversion
  Oral Anticoagulant: warfarin, dabigatran etexilate, rivaroxaban, apixaban, edoxaban usage
Arm/Group | Transesophageal Echocardiography Group | Oral Anticoagulation Group
All-Cause Mortality (participants affected / at risk) | 3/56 | 2/56
Serious Adverse Events (participants affected / at risk) | 9/56 | 10/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transesophageal Echocardiography Group (N=56) | Oral Anticoagulation Group (N=56)
Ischemic stroke-transient ischemic attack (Nervous system disorders) | 4 | 7
Hemorrhagic stroke (Nervous system disorders) | 2 | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 3 | 2

LIMITATIONS AND CAVEATS:
It is a small study. The inclusion criteria were very strict. Patients who required urgent cardioversion, had severe structural heart disease, or conditions that might precipitate atrial fibrillation and those who did not undergo cranial MRI were excluded. Most of the patients had new-onset atrial fibrillation. Therefore the findings of this study cannot be generalized for all atrial fibrillation patients.The evet rates in the both groups were low which decrease the power of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT01924065/Prot_SAP_000.pdf